CLINICAL TRIAL: NCT05889013
Title: A Clinical Study to Gather Data on the Utility of Tests That Are Used to Make a Diagnosis of Primary Ciliary Dyskinesia (PCD)
Brief Title: Utility of PCD Diagnostics to Improve Clinical Care
Acronym: PCD
Status: Recruiting | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: UConn Health (Other)
Responsible Party: Sponsor
Other Study IDs: 23-052-CCMC
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: PCD; nasal nitric oxide testing
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Nasal Nitric Oxide: Participants who are referred by his/her clinician for nasal NO testing and meet the inclusion and exclusion criteria will undergo testing. Clinical information regarding prior diagnostic testing will be collected at time of enrollment. Participants that have a confirmed diagnosis of PCD by genetics or ciliary biopsy at time of study entry
  Interventions: Device: Nasal Nitric Oxide testing

INTERVENTIONS:
Device: Nasal Nitric Oxide testing — Collection of already performed clinical data and nNO testing
  Other Names: nNO testing

SUMMARY:
This cross-sectional and longitudinal observational study is to gather data on the utility of tests that are used to make a diagnosis of primary ciliary dyskinesia (PCD). There is new testing available, called nasal nitric oxide testing, that non-invasively measures nitric oxide levels in the sinus cavity. Individuals with PCD characteristically have low levels, but this testing does not have extensive data from everyday clinical practice. The objective of this proposal is to improve the diagnostic approach to children and adults with clinical concerns for primary ciliary dyskinesia (PCD).

DETAILED DESCRIPTION:
This is an observational study to gather data on the utility of tests that are used to make a diagnosis of primary ciliary dyskinesia (PCD). Participant selection will be on a referral basis for the consideration of a clinical suspicion for PCD. Participants will be identified by pulmonary providers that consider testing for PCD based on the clinical symptoms of the participant. These providers will then refer for enrollment in the study based on the clinical considerations for a diagnosis of PCD. Participants will be consented during the time of testing at the Pulmonary department. Any patient referred by a clinician for concerns for PCD, including those who have had PCD genetics sent, or a ciliary biopsy performed will be enrolled in the study. In addition, any participant who is referred for nasal nitric oxide testing and meets the inclusion and exclusion criteria for this testing, will also need to provide informed consent and be enrolled in the Nasal NO REDCap registry. This equipment is not currently FDA approved or CLIA certified for PCD diagnostic testing and therefore referring clinicians will be informed that the results of this test should not influence clinical decision making regarding the diagnosis of PCD. However, there is growing evidence that this testing has utility as a non-invasive screening tool for PCD and continued data from the general pediatric pulmonary population is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years of age
* Must have two of the following clinical history points:
* Neonatal respiratory distress
* Chronic nasal congestion/runny nose
* Chronic cough
* Situs/laterality defects
* Bronchiectasis
* Ability to provide informed consent or consent of parent/guardian and ass

Exclusion Criteria:

* Recent history of sinus surgery or bloody nose in the past week
* Age < 2 years of age
* Inability to tolerate probe in nose
* Sinusitis or other respiratory exacerbation currently being treated with antibiotics
* Admitted to hospital for respiratory exacerbation (inpatient status)
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by the IRB)
* Any other reason for which the study investigators feel the patient is not a good candidate to complete the testing

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population are ages 2 and up. Participant selection will be on a referral basis for the consideration of a clinical suspicion for PCD. Participants will be identified by pulmonary providers that consider testing for PCD based on the clinical symptoms of the participant. These providers will thenrefer for enrollment in the study based on the clinical considerations for a diagnosis of PCD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Creation of Nasal NO REDCap registry | 2-3 years
  To establish a research registry to characterize the features of individuals that undergo PCD diagnostic testing at Connecticut Children's Medical Center and UCONN.
Evaluation of utility of PCD diagnostic testing | 2-3 years
  To evaluate the utility of PCD diagnostic testing, including potential use of nasal nitric oxide in comparison to genetic testing and ciliary biopsy, in pulmonary practice at Connecticut Children's Medical Center and UCONN.

SECONDARY OUTCOMES:
Refinement and Improvement of PCD Diagnostic Testing | 1-2 years
  To refine and improve current diagnostic processes for PCD diagnosis at CCMC using information gathered from the research registry established through Primary aims 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie S Collins, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Pulmonary Division, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No